CLINICAL TRIAL: NCT02677727
Title: A Study of the Natural History of Cisplatin-Induced Peripheral Neuropathy in Patients With Germ Cell Tumor
Brief Title: Study of Cisplatin-Induced Peripheral Neuropathy in Patients With Germ Cell Tumor
Status: Completed | Type: Observational
Sponsor: Costantine Albany (Other)
Collaborators: Mayo Clinic (Other)
Responsible Party: Sponsor-Investigator, Costantine Albany, Assistant Professor of Medicine, Indiana University School of Medicine
Organization: Indiana University (Other)
Other Study IDs: IUSCC-0502; 1412960547 (Other: Indiana University IRB)
Record Dates: First submitted 2016-02-05; First posted 2016-02-09 (Estimated); Last update posted 2020-09-22 (Actual); Status verified 2020-09

CONDITIONS: Testicular Germ Cell Tumor
Keywords: Cisplatin-based chemotherapy; Chemotherapy-induced peripheral neuropathy
MeSH Terms: conditions — Testicular Germ Cell Tumor

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — DNA to use for future planned evaluations to predict patients at higher risks of developing neuropathy
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: EORTC QLQ-CIPN20 — EORTC QLQ-CIPN20 is a 20-item chemotherapy-induced peripheral neuropathy-specific questionnaire which includes three scales assessing sensory (9 items: #31-36, 39, 40, 48), motor (8 items: #37, 38, 41-45, 49), and autonomic (3 items: #46, 47, 50) symptoms and functioning with each item measured on a 1-4 scale (1 - not at all; 4 - very much).

SUMMARY:
This is a prospective observational study investigating the incidence, characteristics of, and change in chronic neuropathy symptoms related to cisplatin using the EORTC CIPN-20 instrument. Approximately 60 patients will be collected for this study. The duration of this study will be up to 18 months for each patient. This study will complement a current R01 funded trial (Platinum Study) which evaluates the genetic predisposition of chronic neuropathy after 12 months of chemotherapy. However, although the platinum study evaluates a similar patient population, it does not evaluate the natural history of platinum induced neuropathy during active treatment and the first 12 months post chemotherapy. This trial will fill this gap and add to the investigators knowledge for both natural history and genetic predisposition of platinum neurotoxicity.

DETAILED DESCRIPTION:
Primary Objective:

To describe the incidence and characteristics of, and change in, chronic neuropathy symptoms related to cisplatin, using the EORTC CIPN-20 instrument

Procedures:

The EORTC QLQ-CIPN20 questionnaire will be completed on day one of each cycle of chemotherapy, once every three weeks (+/-7 days) and once every 2 months (+/- 30 days) from the last dose of chemotherapy. Patients will be asked to complete the questionnaire in clinic during their routine visits.

As part of this study, a DNA blood sample will be collected and stored with the Indiana Biobank on Day 1 of Cycle 1.

ELIGIBILITY:
Inclusion criteria:

1. 15 years of age or older at the time of informed consent
2. Have a confirmed pathologic and/or by tumor marker diagnosis of testicular or extragonadal germ cell cancer.
3. Provide written informed consent and assent (if applicable).
4. Ability to complete questionnaire(s) in English by themselves or with assistance.
5. Willing to provide a 10 mL blood sample for future DNA testing
6. Planning to receive at least 3 cycles of cisplatin (20 mg/m2/d for 5 days) based chemotherapy.
7. Must agree to continued clinical follow-up at the study cancer center.

Exclusion criteria:

1. Diagnosis (current or previous) of peripheral neuropathy (from diabetes or other causes).
2. Previous exposure to neurotoxic chemotherapy drugs including taxanes, platinum agents, vinca alkaloids, or epothilones.
3. Salvage chemotherapy treatment or bone marrow transplant. Salvage chemotherapy is defined as any treatment after relapse of the disease following initial chemotherapy treatment.

Min Age: 15 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients who are beign treated with cisplatin-based chemotherapy for testicular germ cell tumor
Sampling Method: Non-Probability Sample
Enrollment: 54 (Actual)
Dates: Start 2015-07-01 (Actual); Primary Completion 2020-06-17 (Actual); Study Completion 2020-06-17 (Actual)

PRIMARY OUTCOMES:
Incidence of neuropathy | 18 months
  As measured by cumulative EORTC CIPN-20 scores

SECONDARY OUTCOMES:
Change in neuropathy | 18 months
  As measured by change in EORTC CIPN-20 scores

CONTACTS AND LOCATIONS:
Overall Officials: Costantine Albany, MD, Principal Investigator — Indiana University School of Medicine, Indiana University Simon Cancer Center
Locations (3):
- United States (3):
  - Indiana University Health Hospital, Indianapolis, Indiana
  - Indiana University Health Melvin and Bren Simon Cancer Center, Indianapolis, Indiana
  - Mayo Clinic Department of Medical Oncology, Rochester, Minnesota

REFERENCES:
- [Derived] Albany C, Dockter T, Wolfe E, Le-Rademacher J, Wagner-Johnston N, Einhorn L, Lafky JM, Smith E, Pachman D, Staff N, Ma C, Loprinzi CL, Costello BA. Cisplatin-associated neuropathy characteristics compared with those associated with other neurotoxic chemotherapy agents (Alliance A151724). Support Care Cancer. 2021 Feb;29(2):833-840. doi: 10.1007/s00520-020-05543-5. Epub 2020 Jun 4. PMID 32500206